CLINICAL TRIAL: NCT00495560
Title: A Pilot Study of Priming Before Induction Termination of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26135
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Abortion, Induced; Abortion, Second Trimester
Keywords: induction; abortion; injection, intra-amniotic; misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Addition of misoprostol 25 mcg 12 hours before induction — Misoprostol given buccally the night before induction

SUMMARY:
Induction termination of pregnancy (second trimester abortion) has a median time of 14 hours from the start of medication (misoprostol) to expulsion of the fetus. The objective of this study is to evaluate a method of 'priming' on the length of induction termination of pregnancy. "Priming" refers to the use of medication to ready the cervix and uterus so that the uterus is more sensitive to medication and contracts more effectively, and also refers to softening of the cervix so that there is less resistance to dilation. Priming is used extensively before induction of labor for term pregnancy and is also used extensively before surgical abortion in second trimester. We would like to add priming the evening before induction to the usual treatment and evaluate whether the length of the induction process is shortened. Women are admitted to the hospital in the morning to start misoprostol medication, and unless expulsion occurs within 8-10 hours, need to stay overnight.

The study design is to give the priming dose 12 hours before admission. The outcome of interest is the induction time from the first dose on misoprostol in the hospital to expulsion of the fetus.

This study aims to assess whether the use of misoprostol as a priming agent would be beneficial with women who undergo induction termination of pregnancy.

DETAILED DESCRIPTION:
This is a prospective series. All women enrolled will receive the same treatment. 10 women without prior births and 10 women with prior births will be enrolled. The study design is to give the priming dose 12 hours before admission.

The outcome of interest is the induction time from the first dose on misoprostol in the hospital to expulsion of the fetus.

Inclusion criteria: Women who have requested induction abortion and completed the counseling and consent process for abortion. Women 18 years of age or over. Capable of giving informed consent. Speak English or Spanish Pregnancy 18-23 weeks. No contraindication to misoprostol abortion

Exclusion criteria: Unable to understand and give informed consent. Pregnancy less than 18 weeks or over 23 weeks on the day of enrollment. Ruptured membranes or signs of infection (temperature over 100.6 F,WBC >15K) Fetal demise Multi-fetal pregnancy Contraindication to any of the agents used for misoprostol induction abortion

After women have started the abortion process (completed counseling and consent for abortion, and completed the fetocidal digoxin injection), they will be approached by one of the investigators. The procedures and the consent process will be explained. If they consent, they will be given an envelope which contains 50 mcg of misoprostol (1/2 of a 100 mcg tablet). They will be instructed to place the tablet buccally and hold it in place for 30 minutes, after which it can be swallowed, between 8 and 9 pm that evening.

They will return at 7 am the next morning; the actual induction process starts between 8 and 10 am depending on the bed situation. The reminder of the care is identical to women not in the study and consists of misoprostol 400 every 6 hours. The only step that will be from the current induction process is the administration of the priming dose the night before.

The duration of participation for individuals is up to 48 hours. The study overall will take one year.

Analytic plan:

This is a pilot study to estimate the effect on induction times, and to monitor for any adverse events. This pilot will be the basis of further study.

When the sample size is 19, a two-sided 95.0% confidence interval for a single mean will have an interval that extends no more than 1.5 from the observed mean, assuming that the true standard deviation is 3.25 and that the confidence interval is based on the t statistic. The "typical" mean is 14 hours and the 95% confidence interval around 12.5 hours is 11hours to 14 hours.

The primary outcome is the induction time, the time from start of induction until fetal expulsion. As there are about 80 induction procedures per year, and past studies have enrolled 50-60% of eligible women, it will take approximately 6 months to complete enrollment.

The length of induction will be described and the mean will be contrasted to a typical value (14 hours) . Minor events such as nausea will be tabulated. There will be a sub-analysis of outcome by parity (women without prior births compared to women with prior births). This study is not powered to show differences between these two groups but this information wil be helpful in planning future studies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* able to give informed consent in English or Spanish
* requesting termination of pregnancy
* pregnancy 18-23 weeks of gestation

Exclusion Criteria:

* Unable to understand and give informed consent
* Under 18 years of age
* Pregnancy less than 18 weeks or over 23 weeks on the day of enrollment
* Ruptured membranes or signs of infection (temperature over 100.6 F,WBC >15K)
* Fetal demise, Multi-fetal pregnancy contraindication to misoprostol
* contraindication to misoprostol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Length of time between the start and the finish of the induction | 24 h

SECONDARY OUTCOMES:
incidence of nausea and cramping | 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Nilda L Moreno-Ruiz, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States